CLINICAL TRIAL: NCT06989658
Title: Feasibility and Tolerability Study of Wearing a Miniaturized Smart Contact Lens With Healthy Subjects and Patients With Stargardt's Disease
Brief Title: Feasibility and Tolerability Study of Smart Contact Lens With Healthy Subjects and Patients With Stargardt's Disease
Acronym: RE-SEE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Ecole Nationale Supérieure Mines - Télécom Atlantique Bretagne Pays de la Loire. (Unknown); StreetLab Vision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: P23-01
Record Dates: First submitted 2025-05-06; First posted 2025-05-25 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Stargardt Disease
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Intervention Model Description: We have made the methodological choice of including healthy volunteers first, in order to validate the feasibility and tolerance of the SCL lens in people with healthy eyes.
  If no serious adverse events occur in the first 12 control subjects, we will then be able to begin enrolling patients with Stargardt's disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with Stargardt disease (Experimental): 16 patients with Stargardt's disease, whose visual acuity will be greater than or equal to 20/400e in binocular vision;
  Interventions: Device: SCL miniaturized scleral lens positioning
- Healthy volunteers (Active Comparator): 16 healthy volunteers, sighted controls with visual acuity of at least 10/10th in binocular vision.
  Interventions: Device: SCL miniaturized scleral lens positioning

INTERVENTIONS:
Device: SCL miniaturized scleral lens positioning — 1. Experimental evaluation:
     1. TESTs withSCL system
        * Before positioning the SCL lens: slit lamp examination
        * After positioning the SCL lens: slit-lamp examination
        * Tests performed on projected screen.
     2. Tests with a conventional oculometer: tests performed on a projected screen.
  2. Ophthalmological assessment:
     1. slit lamp examination
     2. An end-of-study follow-up phone call.

SUMMARY:
Oculometry is becoming increasingly popular in fields such as enhanced reality and healthcare, but remains limited by complex devices that are poorly adapted to the needs of users, particularly the visually impaired. This research proposes to explore a smart contact lens (SCL)-based system to overcome these limitations, particularly for people with central visual deficits such as Stargardt's disease.

DETAILED DESCRIPTION:
Eye tracking is becoming increasingly important in fields such as augmented reality such as augmented reality, virtual reality and healthcare (orthoptic rehabilitation), but is still limited by complex measurement methods that meet user needs.

In this context, the proposed research aims to study the feasibility of a system based on a smart contact lens that overcomes several overcome many of the limitations of current oculometers (sensitivity to environmental sensors, size, performance, etc.) and even more so when used by visually impaired people suffering from central vision deficits central vision deficit such as Stargardt's disease. Whether to eccentric fixation or to transmit relevant information about the environment relevant information about their environment, it is necessary to know direction of gaze. Unfortunately, current solutions are not always compatible with the difficulties faced by visually impaired and the SCL system could be a viable and effective solution.

ELIGIBILITY:
Inclusion Criteria:

Patients with Stargardt disease

* Age: 18 - 70 ;
* Juvenile form of Stargardt's disease manifested by decreased visual acuity;
* Visual acuity greater than or equal to 20/400 in binocular vision;
* MMSE score without visual item ≥ 20/25 ;
* Eyes whose palpebral opening and ocular surface and its appendages allow the wearing of a scleral lens;
* Sufficient knowledge of the French language.
* Ability to give express, free and informed consent in person, after having received adequate information;
* Ability to comply with protocol requirements;
* Person covered by Health Insurance.

Healthy volunteers:

* Age: 18 - 70 years;
* Age- and sex-matched healthy volunteers to subjects with Stargardt's disease (± 5 years);
* MMSE score with visual items ≥ 25/30 ;
* Eyes with palpebral opening and ocular surface and appendages suitable for scleral lens wear;
* Visual acuity of at least 10/10 in binocular vision;
* Sufficient knowledge of the French language;
* Ability to give personal, express, written, free and informed consent after receiving adequate information ;
* Ability to comply with protocol requirements;
* Person covered by Health Insurance.

Exclusion Criteria:

For all participantsPersons referred to in articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons : pregnant women, parturients, nursing mothers, persons deprived of liberty by judicial or administrative decision, minors, and persons subject to a legal protection measure: guardianship or curatorship);

* Participants with neurodegenerative diseases or any other disease that could interfere with the planned evaluations during this study;
* Participants with ophthalmological diseases other than Stargardt's disease;
* Participants with a history of cleft palate, corneal infection, irregular cornea (such as keratoconus) and severe dry eye syndrome as determined by the ophthalmologist;
* Participants allergic or sensitive to methyl acrylic poly methacrylate (PMMA) or to any of the components of the Re-See lens;
* Participants allergic to tropicamide, atropine or its derivatives
* Participants at risk of angle-closure glaucoma;
* Participants allergic to sodium fluorescein;
* Suspicion of transmissible spongiform encephalopathy;
* Medications that may cause motor, visual or cognitive disorders (neuroleptics, etc.) or that may interfere with study evaluations;
* Participation in another clinical trial that could interfere with the present study;
* Inability to follow instructions or read. ☞Wearing glasses or contact lenses is not a non inclusion criterion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence rate of adverse events, unexpected adverse events or serious adverse events | 45 days
  Ophthalmological consultation (including slit-lamp corneal examination) and subject interrogation. Each reported event will be analyzed to monitor its evolution (resolution or not, necessary treatments...) and to estimate the imputation with the wearing of the LCS lens.
Ergonomics evaluation | 45 days
  To evaluate the ergonomics: comfort, acceptability and usefulness of the SCL lens with subjects suffering from central vision deficit (Stargardt's disease) and healthy control subjects, we will use the satisfaction questionnaire we have specially designed. Analysis of the results of the close-ended and semi-open-ended questions will enable us to answer this question.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle AUDO, MD, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France